CLINICAL TRIAL: NCT00760708
Title: Circulating Adenosine Levels Before and After Intravenous (IV) Persantine
Status: Terminated | Type: Observational
Why Stopped: Persantine is no longer being used at UCHC for pharmacological stress testing
Sponsor: UConn Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bruce Liang, Professor of Medicine, Director Pat and Jim Calhoun Cardiovascular Center, UConn Health
Other Study IDs: 02-115-1; Proposal Number 04156012; Award NumberW81XWH-05-1-0060
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Ischemia; Coronary Disease
Keywords: nucleosides; neurotransmitter; myocardial ischemia; Adenosine
MeSH Terms: conditions — Ischemia; Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- undergoing persantine stress test

SUMMARY:
Persantine is a drug that is routinely used to determine blood flow to the heart in the diagnosis of coronary heart disease. Persantine causes an increase in the adenosine level in the blood. Adenosine is a naturally occurring substance in the body that can increase blood flow. Adenosine is normally removed from the bloodstream by an adenosine transporter, which is a protein that takes up adenosine from the blood into cells. The increase in adenosine levels in the blood is variable, and the cause for this variability is unknown. A mutation for this transporter gene may contribute to this variability, and may alter its function. Thus, the purpose of this study is to determine the relationship between the mutation and the transporter function.

DETAILED DESCRIPTION:
Objectives:

The overall goal of this proposal is to develop methods to achieve heart and vascular protection from ischemia and thus improve soldier's performance in adverse environment. The major hypothesis is that new approach and method can be developed to enhance resistance to stress-induced circulatory insufficiency and myocardial ischemia. The goals here are to determine whether a decreased adenosine transporter function is associated with a reduced physiological responsiveness to the vasculo-protective drug persantine using two in vitro endpoints: the ability of persantine 1) to inhibit platelet aggregation and 2) to inhibit [3H] uridine uptake. Both are endpoints that indicate physiological responsiveness. Both relate directly to the cardiovascular protective effects of , that is, persantine the availability of extracellular adenosine level and the anti-platelet property. Specifically, the relationship between circulating adenosine increase to persantine in vivo and blockade of radio-labeled uridine uptake by erythrocytes and of platelet aggregation by the drug in vitro will be determined. These investigations will recruit subjects undergoing persantine stress testing in the Nuclear Cardiology Laboratory.

Scientific Background and Significance:

Development of methods to protect from skeletal and cardiovascular insufficiency is the main objective of the current research. Adenosine is a potent cyto-protective hormone released during ischemia. The goal of this clinical research project are to test the presence of genetic polymorphisms in the adenosine transporter gene and to determine whether it is associated with an altered persantine responsiveness. The hypothesis is that some or all of these polymorphisms are associated with a decreased responsiveness to persantine and that increasing the dose of persantine will overcome the relative non-response.

Specific Evaluations:

-Persantine Administration: Persantine will be administered after baseline evaluation with intravenous dose (0.56 mg/kg) over 5 minutes.

-Adenosine levels: Adenosine levels will be measured at baseline, and 2 minutes after the persantine dose. We have recently modified and adapted a method to measure nanomolar concentration of adenosine in human blood.

-Adenosine transporter function: The transporter function will be determined by the ability of persantine to inhibit erythrocyte uptake of radio-labeled uridine in vitro.

- Anti-platelet effect of persantine: The platelet aggregation response to persantine will be determined via whole blood aggregometry in vitro where the ex vivo platelet response to the drug can be quantified.

Preliminary Studies:

Preliminary data showed that two non-synonymous single nucleotide polymorphisms occurring at a frequency of 3-4% exist in the persantine-binding regions of the adenosine transporter gene. The goal of the present study is to determine the functional significance of these polymorphisms by testing the association of these polymorphisms with the ability of persantine to inhibit uridine (uridine uses the same transporter) uptake and platelet aggregation. These represent the in vitro functional endpoints in the subjects with the polymorphism. The investigators will also study the association of these polymorphisms with any clinical characteristics such as the incidence of MI, acute coronary syndrome, coronary bypass or stenting procedures. Since this is NOT an interventional study, these are not considered clinical outcomes or endpoints in the traditional sense when an intervention is carried out. These are considered clinical characteristics or phenotypes that associate with the genotype of polymorphisms. Primary and secondary outcomes and endpoints: The goal of the present study is to determine the functional significance of these polymorphisms by testing the association of these polymorphisms with the ability of persantine to inhibit uridine (uridine uses the same transporter) uptake and platelet aggregation. These represent the in vitro functional endpoints in the subjects with the polymorphism. The investigators will also study the association of these polymorphisms with any clinical characteristics such as the incidence of MI, acute coronary syndrome, coronary bypass or stenting procedures. Since this is NOT an interventional study, these are not considered clinical outcomes or endpoints in the traditional sense when an intervention is carried out. These are considered clinical characteristics or phenotypes that associate with the genotype of polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with or without coronary artery disease undergoing a Persantine nuclear stress test

Exclusion Criteria:

* Oral persantine use within 24 hours
* Second or third degree AV block, or sick sinus syndrome without a functioning pacemaker
* Active asthma or bronchospasm
* Those with end-stage liver disease such as cirrhosis or active hepatitis such as > 5 fold liver enzyme elevation will not be included
* Anemia (Hct < 30)
* Myocardial infarction within 30 days
* Severe left ventricular dysfunction (EF < 30%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing a Persantine nuclear stress test for medically-indicated reasons. There are no control subjects.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine functional significance and association of these polymorphisms with the ability of persantine to inhibit uridine (uridine uses the same transporter) uptake and platelet aggregation. | 24 hours

SECONDARY OUTCOMES:
Investigators will study the association of these polymorphisms with any clinical characteristics such as the incidence of MI, acute coronary syndrome, coronary bypass or stenting procedures. These clinical outcomes are considered secondary endpoints. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Liang, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States